CLINICAL TRIAL: NCT02737891
Title: A Double-blind, Randomized, Placebo-controlled, Multiple-dose, Two-center, Safety and Efficacy Study of Co-administration of Tesofensine/Metoprolol Treatment in Subjects With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Safety and Efficacy Study of Tesofensine/Metoprolol Treatment in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Saniona (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TM001
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tesofensine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tesofensine/Metoprolol (Experimental): Oral tablets Tesofensine/Metoprolol
  Interventions: Drug: Tesofensine/Metoprolol
- Placebo (Placebo Comparator): Placebo tablets matching oral Tesofensine/Metoprolol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tesofensine/Metoprolol — Tesofensine 0.5 mg + Metoprolol 100 mg
  Other Names: Tesofensine; Metoprolol
  Arms: Tesofensine/Metoprolol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Safety and Efficacy Study of Tesofensine/Metoprolol Treatment in Subjects With Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, multiple-dose, two-center, safety and efficacy study of co-administration of tesofensine/metoprolol treatment in subjects with T2DM. Study medication will be administered for ninety (90) days (+2 days after the final assessments with half-dose of metoprolol). Following all baseline assessments, eligible subjects will be randomly assigned to one of the two arms (1:1).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Confirmed diagnosis of T2DM
3. 18-70 years of age
4. HbA1c ≥7.0%

Exclusion Criteria:

1. Hypersensitivity to tesofensine/metoprolol
2. Heart failure class II or greater according to the New York Heart Association (NYHA) or decompensated heart failure
3. History of myocardial infarction or stroke within 12 months prior to enrolment
4. History of coronary revascularisation or angioplasty in the last 12 months prior to enrolment
5. Patients reporting angina in the last 6 months prior to enrolment
6. Treatment with insulin and/or other injectable anti-diabetic medications, or TZDs
7. Any clinically significant cardiac arrhythmia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Drejer, PhD, Study Director — Saniona
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablets matching oral Tesofensine/Metoprolol
  Placebo
Period: Overall Study
Arm/Group | Tesofensine/Metoprolol | Placebo
Started | 30 | 30
Completed | 30 | 28
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tesofensine/Metoprolol | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (7) | 64 (5) | 64 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 21
  Male | 15 | 24 | 39

OUTCOME MEASURES:

1. Primary Outcome: Effects of Co-administration of Tesofensine/Metoprolol Treatment vs. Placebo on 24-hour Mean Heart Rate
Description: 24-hour heart rate monitoring was based on telemetry measurements at baseline (Day -1 to 1, V2) and at the end of treatment (Day 90 to 91, V10). The heart rate was measured every minute and the mean was recorded for every hour.
Time Frame: Baseline to Day 90
Measure: Mean (Standard Deviation); unit: beats per minutes (BPM)
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 30 | 30
beats per minutes (BPM) | 67 (7) | 70 (9)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol vs Placebo; The analysis was based on a parametric model, i.e. compared between treatment arms by means of an analysis of covariance (ANCOVA) model (proc MIXED) using change from baseline to the end of treatment as dependent variable, treatment and study site as fixed effects and the value from baseline as covariate. The residual errors were assumed independent and identically distributed (i.i.d.) and normally distributed; Test type: Superiority; p = 0.004, ANCOVA — Two-sided p-value for test of no difference from 0; Mean Difference (Net) = -3.8, 95% CI 2-sided [-6.36 to -1.29]

2. Secondary Outcome: Change From Baseline to End of Treatment in HbA1c
Description: HbA1c was measured from blood samples collected at baseline (Day 1, V2) and at the end of treatment (Day 90, V10). Additional HbA1c measurements were done during various visits (V6, V8 and V12).
Time Frame: Baseline to Day 90
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 30 | 30
percentage of HbA1c | 7.3 (0.6) | 7.4 (0.7)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.724, ANCOVA — Two-sided p-value for test of no difference from 0; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.23 to 0.33]

3. Secondary Outcome: Change From Baseline to End of Treatment in Body Weight
Description: Change in kg body weight measured from baseline to day 90
Time Frame: Baseline to Day 90
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Tesofensine/Metoprolol | Placebo
Number analyzed (Participants) | 30 | 30
kg | -3.5 (19.9) | -0.3 (12.9)
Statistical Analysis 1: Comparison: Tesofensine/Metoprolol vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Two-sided p-value for test of no difference from 0; Mean Difference (Net) = -3.5, 95% CI 2-sided [-4.65 to -2.30]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from baseline to D90. 90days. • Change from baseline to end of treatment
Arm/Group | Tesofensine/Metoprolol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/30
Other Adverse Events (participants affected / at risk) | 20/30 | 12/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tesofensine/Metoprolol (N=30) | Placebo (N=30)
cholelithiasis (Metabolism and nutrition disorders) | 0 | 1 — One not treatment-emergent SAE; placebo arm,moderate intensity; rated not related to study drug; outcome recovered/resolved.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tesofensine/Metoprolol (N=30) | Placebo (N=30)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (11) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Asthenia (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 3 (3) | 0 (0)
Hot flush (General disorders) | 1 (1) | 0 (0)
Hyperhidrosis (General disorders) | 6 (6) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Application site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye burns (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Oedema peripheral (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (12) | 1 (1)
Headache (Nervous system disorders) | 5 (10) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Disturbance in attention (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 3 (3) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Herpes simplex (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail injury (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dental implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT02737891/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT02737891/SAP_001.pdf